CLINICAL TRIAL: NCT03595982
Title: Is Procardia XL 60 mg Q Daily Equivalent to 30 mg XL Given Twice Daily?
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Melissa Chu Lam, Maternal Fetal Medicine Fellow, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 18-0959
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Results first posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Hypertension in Pregnancy; Hypertension in Postpartum
Keywords: chronic hypertension; postpartum hypertension; preeclampsia; treatment; Procardia XL
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia | interventions — Nifedipine

STUDY DESIGN:
Intervention Model Description: Depending on the group the person gets randomized into they will receive 60 mg of nifedipine at 0h vs 30 mg of nifedipine at 0h followed by 30 mg extra at 12h, These medications will be administered by a nurse or physician on the floor.
  After 12h and at the end of the 24h (plus or minus 30 min) a blood sample (2cc) with be obtained and sent to Mount Sinai Hospital to determine serum Procardia levels. This blood samples will be stored until this research study is finished and will be disposed after. A total of 20cc of blood will be obtained from each patient.
  Also the patient will take a survey of side effects of the BP medication. BPs will be measured Q 4h and documented at 0h, 4h, 8h, 12h, 16h, 20h and 24h (plus or minus 30 min)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Procardia XL 30 mg (Experimental): Procardia XL 30 mg XL Q 12h - When a patient's BP is persistently elevated after a dose of 30 mg of Procardia XL, the dose is increased to 60 mg Procardia XL divided in 2 doses of 30 mg given 12h apart.
  Interventions: Drug: Procardia XL 30Mg
- Procardia XL 60 mg (Active Comparator): Procardia XL 60 mg Q 24h - When a patient's BP is persistently elevated after a dose of 30 mg of Procardia XL, the dose is increased to 60 mg Procardia given once a day.
  Interventions: Drug: Procardia XL 60Mg

INTERVENTIONS:
Drug: Procardia XL 30Mg — Procardia XL 30 mg XL Q 12h
  Arms: Procardia XL 30 mg
Drug: Procardia XL 60Mg — Procardia XL 60 mg Q 24h
  Arms: Procardia XL 60 mg

SUMMARY:
Antihypertensive therapy has been used in pregnant patients antepartum to improve blood pressure (BP) elevation in cases of chronic hypertension, and postpartum for persistent hypertension after delivery in cases of gestational hypertension and preeclampsia, as well as for management of chronic hypertension.

There is limited evidence regarding the precise BP level at which antihypertensive therapy is indicated during pregnancy for chronic hypertension. Treatment has been suggested in pregnant patients when systolic BP is ≥ 160 mmHg and at a lower diastolic BP threshold of 105 mm Hg, however some providers may initiate therapy at systolic BPs ≥ 150 mmHg.

Nifedipine is a peripheral arterial vasodilator and an ideal first line antihypertensive agent due to its low maternal side-effect profile. It has been proven to be safe in pregnancy. Conventional nifedipine can be started at 10 mg twice daily with a maximum dose of 120 mg/d, but frequently extended release tablets are preferred due to steady blood pressure control with once daily administration.

It is frequently used however as a twice daily dosing as many providers have noticed an increase in the BPs 12-24h from administration. Twice daily dosing might produce overlapping profiles that prevent elevation of BP at the time of the next administration and breakthrough elevations throughout the day in pregnant women.

The aim of this study is to investigate the mean plasma levels and standard deviations of Procardia at 24h after Procardia XL is administered as a 60 mg daily dose and the mean plasma levels after it is given as a 30 mg twice-daily dose. This will be a pilot study for a future randomized control trial that will allow the researchers to determine whether 60 mg daily of Procardia XL is equivalent to 30 mg twice daily. Secondary outcome will be effective control of BP throughout the day (0h, 4h, 8h, 12h, 16h, 20h and 24h) defined as BPs below 160/105 as well as side effects of nifedipine as reported by patients.

DETAILED DESCRIPTION:
There is limited evidence regarding the precise BP level at which antihypertensive therapy is indicated during pregnancy for chronic hypertension. Given the limitations of data as well as higher likelihood of outpatient therapy with less frequent blood pressure monitoring, treatment has been suggested in pregnant patients when systolic BP is ≥ 160 mmHg and at a lower diastolic BP threshold of 105 mm Hg , however some providers may initiate therapy at systolic BPs ≥ 150 mmHg.

Antihypertensive therapy has not been shown to improve fetal condition or to prevent preeclampsia. However, such therapy controls acceleration of BP, reduces antepartum hospitalization due to severe hypertension and should help prevent maternal complications from uncontrolled hypertension such as cardiovascular (congestive heart failure and myocardial ischemia), renal (renal injury or failure), or cerebrovascular (ischemic or hemorrhagic stroke) damage.

Drugs such as methyldopa, labetalol, and nifedipine in many occasions are used as first line agents for control of hypertension in pregnancy.

Calcium channel blockers are a class of drugs that have not been extensively studied in pregnant women with chronic hypertension, however they are still considered standard of care for treatment of elevated BPs during pregnancy and after delivery. Small amounts have been shown to cross the placenta, however to date no known association with birth defects have been found with reassuring long term follow-up of babies up to 1.5 years. It is not associated with adverse perinatal outcomes and furthermore, nifedipine does not appear to adversely affect uterine or umbilical blood flow.

Nifedipine is a peripheral arterial vasodilator and an ideal first line antihypertensive agent due to its low maternal side-effect profile. Conventional nifedipine can be started at 10 mg twice daily with a maximum dose of 120 mg/d, but frequently extended release tablets are preferred due to steady blood pressure control with once daily administration. The extended release tablet consists of a semipermeable membrane surrounding an osmotically active drug core and has been designed to provide nifedipine an approximately constant rate over 24h.

ELIGIBILITY:
Inclusion Criteria:

* Antepartum or postpartum patients between the age of 18-55 requiring 60 mg of Procardia XL to control elevated blood pressures secondary to preeclampsia, gestational hypertension, or chronic hypertension.

Exclusion Criteria:

* All patients receiving other antihypertensive medication
* All patients with a contraindication to nifedipine: Hypersensitivity to nifedipine or other calcium -channel blocker, cardiogenic shock, concomitant administration with strong CYP34A inducers (rifampin, rifabutin, phenobarbital, phenytoin, carbamazepine, St Johns Wort) → significantly reduces nifedipine efficacy, impaired liver function→? Patients with hepatic impairment (liver cirrhosis) have a longer disposition half-life and higher bioavailability of nifedipine than healthy volunteers
* Patients over the age of 55

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 5 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa T Chu Lam, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Manninen AK, Juhakoski A. Nifedipine concentrations in maternal and umbilical serum, amniotic fluid, breast milk and urine of mothers and offspring. Int J Clin Pharmacol Res. 1991;11(5):231-6. PMID 1814844
- [Background] Clement S, Bowen-Wright H. Twenty-four hour action of insulin glargine (Lantus) may be too short for once-daily dosing: a case report. Diabetes Care. 2002 Aug;25(8):1479-80. doi: 10.2337/diacare.25.8.1479-a. No abstract available. PMID 12145255
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- [Background] Berghella, V., Maternal-Fetal Evidence Based Guideline. Third Edition ed. Series in Maternal-Fetal Medicine, ed. G.C.D.R.a.D. Maulik. 2017, Boca Raton, FL: Taylor ans Francis Group, LLC.
- [Background] Procardia XL [package insent}. Pfizer Labs, New York, NY, 2016. Available from: http://labeling.pfizer.com/ShowLabeling.aspx?id=542. Accessed Novemeber 12, 2017.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Procardia XL 30 mg | Procardia XL 60 mg
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Procardia XL 30 mg | Procardia XL 60 mg | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (9) | 35 (0) | 38 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Procardia Plasma Level
Description: Procardia plasma level at 24 hours after Procardia administration
Time Frame: at 24 hours
Population: Data not collected
Arm/Group | Procardia XL 30 mg | Procardia XL 60 mg
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Blood Pressure (Systolic/Diastolic)
Description: Blood pressure reading
Time Frame: up to 24 hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Procardia XL 30 mg | Procardia XL 60 mg
Number analyzed (Participants) | 3 | 2
mmHg
  Systolic | 155 (14) | 146 (2)
  Diastolic | 92 (10) | 84 (5)

3. Secondary Outcome: Survey of Side Effects
Description: Survey to assess Frequency of side effects of nifedipine including peripheral edema (most common side effect, dose related), flushing, headache, dizziness, fatigue, constipation, nausea, and muscle cramps.
Time Frame: up to 24 hours
Measure: Number; unit: events
Arm/Group | Procardia XL 30 mg | Procardia XL 60 mg
Number analyzed (Participants) | 3 | 2
events | 1 | 2

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Procardia XL 30 mg | Procardia XL 60 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 1/3 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Procardia XL 30 mg (N=3) | Procardia XL 60 mg (N=2)
Headache (Nervous system disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT03595982/Prot_SAP_000.pdf